CLINICAL TRIAL: NCT06520553
Title: A Double-micro-tracer Human Absorption, Distribution, Metabolism and Excretion (hADME) and Absolute Bioavailability Trial After a Single Oral Dose of BI 1569912 (C-14) and a Single, Concomitant, Intravenous Micro-dose of BI 1569912 (C-13) in Healthy Male Subjects (a Phase I, Open-label, Non-randomised, Single-dose, Fixed-sequence Trial)
Brief Title: A Study in Healthy Men to Test How BI 1569912 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1447-0010; 2023-510464-12-00 (Registry Identifier: CTIS); U1111-1302-4229 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 1569912 (C-14) followed by BI 1569912 (C-13) (Experimental): BI 1569912 (C-14) = [test treatment, T] BI 1569912 (C-13) = [reference treatment, R]
  Interventions: Drug: BI 1569912 (C-14); Drug: BI 1569912 (C-13)

INTERVENTIONS:
Drug: BI 1569912 (C-14) — unlabelled BI 1569912 mixed with [14C]- labelled BI 1569912
Drug: BI 1569912 (C-13) — [13C]- labelled BI 1569912

SUMMARY:
The main objectives of this trial are:

* To investigate basic pharmacokinetics of BI 1569912 and total radioactivity, including mass balance, excretion pathways and metabolism following oral administration of BI 1569912 (C-14) to healthy male subjects (test treatment, T).
* To investigate the absolute bioavailability of BI 1569912 as single oral solution dose, using a single, concomitant intravenous micro-tracer administration of BI 1569912 (C-13) (reference treatment, R)

ELIGIBILITY:
Inclusion Criteria :

Subjects will only be included in the trial if they meet the following criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m 2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria :

Subjects will not be allowed to participate, if any of the following general criteria apply:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 40 to 100 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) after repeated measurements
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery for [ 14 C]- radioactivity in urine after oral administration of BI 1569912 (C-14): fe urine,0-tz (fraction excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to Day 14.
Mass balance recovery for [ 14 C]- radioactivity in faeces after administration of BI 1569912 (C-14): fe faeces,0-tz (fraction excreted in faeces as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to Day 14.
Mass balance recovery for [14C]- radioactivity in urine and faeces after oral administration of BI 1569912 (C-14): Sum of feurine,0-tz and fefaeces,0-tz (total recovery of [14C]-radioactivity) | up to Day 14.
AUC0-∞ (area under the concentration-time curve over the time interval from 0 extrapolated to infinity in plasma) of BI 1569912 after a single oral administration of BI 1569912 (C-14) | up to Day 13.
AUC0-∞ (area under the concentration-time curve over the time interval from 0 extrapolated to infinity in plasma) of [ 13 C] BI 1569912 after a single intravenous infusion of BI 1569912 (C-13) | up to Day 6.

SECONDARY OUTCOMES:
Cmax (maximum measured concentration in plasma) of BI 1569912 after a single oral administration of BI 1569912 (C-14) | up to Day 13.
AUC0-tz (area under the concentration-time curve over the time interval from 0 to the last quantifiable time point in plasma) of BI 1569912 after a single oral administration of BI 1569912 (C-14) | up to Day 13.
Cmax (maximum measured concentration in plasma) of [ 14 C]-radioactivity after a single oral administration of BI 1569912 (C-14) | up to Day 13.
AUC0-tz (area under the concentration-time curve over the time interval from 0 to the last quantifiable time point in plasma) of [ 14 C]-radioactivity after a single oral administration of BI 1569912 (C-14) | up to Day 13.
Cmax of [ 13 C] BI 1569912 after a single intravenous administration of BI 1569912 (C- 13) | up to Day 6.
AUC0-tz of [ 13 C] BI 1569912 after a single intravenous administration of BI 1569912 (C-13) | up to Day 6.

CONTACTS AND LOCATIONS:
Locations (1):
- ICON-Groningen-62040, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com